CLINICAL TRIAL: NCT06900738
Title: A Study to Evaluate Non-invasive Measurements of the Inflammatory Status in Patients with IBD
Acronym: VERSATILE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: NimBio (Unknown)
Responsible Party: Principal Investigator, Marc Ferrante, Prof. dr. Marc Ferrante, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VERSATILE
Record Dates: First submitted 2025-03-14; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Bowel Disease (IBD); Ulcerative Colitis (UC); Crohn Disease (CD)
Keywords: inflammatory biomarker
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — Photoplethysmography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IBD patients with inflammometer (Other): blood samples, stool samples, questionnaires and inflammometer measurements
  Interventions: Device: Inflammometer

INTERVENTIONS:
Device: Inflammometer — Patients wear an inflammometer for Photoplethysmography measurements.
  Other Names: inflammatory biomarkers; Photoplethysmography

SUMMARY:
Patients with IBD, including both Crohn's disease and ulcerative colitis, require accurate monitoring of intestinal inflammation for optimal follow-up and treatment. Traditional markers like C-reactive protein (CRP) and faecal calprotectin are useful but are either invasive or disliked by patients and a proper continuous monitoring is not feasible with fragmented biomarker information.

The NimBio technology provides support for the clinicians who are managing IBD patients' care based on a wearable technology that allows tracking responsiveness of blood flow properties (also called hemorheology) to inflammatory processes. NimBio's technology analyses blood flow properties using photoplethysmography (PPG), an optical signal, which detects blood flow changes in the microvascular bed of tissues. The PPG signal is obtained from a commercially available wearable (bracelet) which is convenient for the patients. Based on the impact of inflammation on parameters influencing hemorheology (mainly blood vessel stiffness, blood viscosity and red blood cell aggregation) and the fact that the PPG signal mirrors blood flow characteristics, PPG measurements are associated with changes in inflammatory biomarkers and therefore correlate with disease activity.

This offers a possibility for continuous, non-invasive monitoring of inflammation. The study aims to further validate the NimBio Inflammometer and its value for monitoring inflammatory changes and dynamics in patients with IBD at the University Hospitals Leuven.

DETAILED DESCRIPTION:
Patients with IBD, including both Crohn's disease and ulcerative colitis, require accurate monitoring of intestinal inflammation for optimal follow-up and treatment. Traditional markers like C-reactive protein (CRP) and faecal calprotectin are useful but are either invasive or disliked by patients and a proper continuous monitoring is not feasible with fragmented biomarker information.

The NimBio technology provides support for the clinicians who are managing IBD patients' care based on a wearable technology that allows tracking responsiveness of blood flow properties (also called hemorheology) to inflammatory processes. NimBio's technology analyses blood flow properties using photoplethysmography (PPG), an optical signal, which detects blood flow changes in the microvascular bed of tissues. The PPG signal is obtained from a commercially available wearable (bracelet) which is convenient for the patients. Based on the impact of inflammation on parameters influencing hemorheology (mainly blood vessel stiffness, blood viscosity and red blood cell aggregation) and the fact that the PPG signal mirrors blood flow characteristics, PPG measurements are associated with changes in inflammatory biomarkers and therefore correlate with disease activity.

This offers a possibility for continuous, non-invasive monitoring of inflammation. The study aims to further validate the NimBio Inflammometer and its value for monitoring inflammatory changes and dynamics in patients with IBD at the University Hospitals Leuven

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. At least 18 years of age at the time of signing the Informed Consent Form (ICF)
3. Diagnosis of IBD (Crohn's disease or ulcerative colitis) or IBDU
4. Hospitalized or ambulatory patients with active IBD defined as:

   1. HBI ≥ 5, or PMS score ≥3, and
   2. Faecal Calprotectin ≥200 μg/g or CRP > 10 mg/ml, and
   3. Access to iOS or Android-based smartphone with internet access
5. Ambulatory patients would be recruited to the study with a gender ratio that will not deviate from a 40:60 ratio in favor of either gender

Exclusion Criteria:

1. Pregnancy
2. Allergy to steel or elastomer/rubber
3. Using a pacemaker, implantable cardiac defibrillator, neurostimulator, or other electronic medical equipment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of the the PPG signal with any dynamic biomarker | 6 months
  Correlation of the inflammatory dynamics (trajectory) as measured by NimBio's technology with any dynamic biomarker in the IBD patient population

SECONDARY OUTCOMES:
Correlation of the PPG signal with the patient inflammatory status | 6 months
  Correlation of the inflammatory dynamics as measured by NimBio's technology with the patient inflammatory status as defined by any dynamic biomarker as compared to each individual biomarker in the overall IBD patient population.
Classification of the inflammatory status based on the PPG signal | 6 months
  Classification of the inflammatory status as inflamed vs non-inflamed based on NimBio's technology as defined by increase of 1.5-fold over the upper normal limit
Correlation of the inflammatory trajectory with the patient's inflammatory status | 6 months
  Correlation of the inflammatory trajectory as defined by NimBio's technology with the patient's inflammatory status as assessed by HBI, PRO-2, PMS and SCCAI
Classification of the inflammatory status compared to the clinical disease activity | 6 months
  Classification of the inflammatory status as inflamed vs non-inflamed based on NimBio's technology compared to the clinical disease activity measured by disease activity questionnaires (where inflammation is defined as HBI> 5 and PMS>3).
Time of NimBio's indication of a change in the inflammatory status | 6 months
  The time of NimBio's indication of a change in the inflammatory status compared with the time of change in the clinical disease score or a physician instructed treatment modification
Assessment of physiological parameters | 6 months
  Assessment of physiological parameters such as pulse rate, as measured by non-invasive measurements
Assessment of patient satisfaction | 6 months
  Assessment of patient satisfaction about the wearable with PREM questionnaire
Assessment of the correlation between the inflammatory status and disease activity | 6 months
  Assessment of the correlation between the inflammatory status determined by NimBio's technology and disease activity as measured by endoscopy
The effect of the integration of physiological parameters into NimBio's algorithm | 6 months
  The effect of the integration of physiological parameters such as pulse rate into NimBio's algorithm as compared to at least one inflammatory biomarker reflecting the patient's inflammatory status

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Leuven, Belgium